CLINICAL TRIAL: NCT05472545
Title: Dyadic Neurofeedback for Development of Healthy Emotion Regulation in Youth
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oklahoma State University Center for Health Sciences (Other)
Responsible Party: Principal Investigator, Kara Kerr, Assistant Professor, Oklahoma State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2022029-Hardesty
Record Dates: First submitted 2022-07-21; First posted 2022-07-25 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Emotional Regulation
MeSH Terms: conditions — Emotional Regulation | interventions — Neurofeedback

STUDY DESIGN:
Masking Description: Dyads will be randomly assigned to the experimental or control condition. This study cannot have true masking, as participants in the experimental group will know they are receiving neurofeedback. The control group will not be informed of the existence of the neurofeedback condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Neurofeedback Group (Experimental): Mothers of adolescent participants will view real-time fMRI neurofeedback representing activity in their daughter's anterior insula during an emotion discussion task. Activity will be presented as a colored bar of moving height, and mothers will be instructed to attempt to downregulate the activity through what they say to their daughter.
  Interventions: Behavioral: Neurofeedback
- Control Group (No Intervention): The paradigm for the control condition will be identical to that of the experimental condition except that no neurofeedback will be presented. Participants in the control group will be told that we would like to see if the mother can regulate her daughter's brain activity through supportive statements.

INTERVENTIONS:
Behavioral: Neurofeedback — Real-time functional magnetic resonance imaging dyadic neurofeedback
  Arms: Neurofeedback Group

SUMMARY:
This study will examine the effect of a real-time functional magnetic resonance imaging (fMRI) dyadic neurofeedback protocol with mothers and their adolescent daughters. Mothers in the experimental condition will view a moving bar showing their daughters' brain activity on a computer screen while talking to their daughters.

DETAILED DESCRIPTION:
Adolescents with a family history of adverse childhood experiences (ACEs) are at heightened risk for depression and other mental health problems related to poor emotion regulation (ER). The proposed study will test the efficacy of a real-time fMRI dyadic neurofeedback (DNF) protocol to promote healthy ER-related neurodevelopment in female adolescents with a maternal history of ACEs. The proposed study will use DNF to provide neurofeedback from the adolescent's anterior insular cortex (aIC) to the adolescent's mother as the mother and adolescent engage in an emotion discussion task together. Parents and adolescents (n=35 active DNF; n=35 control) will communicate via microphones and noise-canceling headphones while the adolescent is undergoing fMRI scanning. Specific aims of the current study are to determine: 1) the effects of aIC DNF on the developing ER network in adolescents with a history of maternal ACEs, 2) associations between parenting practices during DNF and reduced adolescent aIC activation, and 3) longitudinal effects of aIC DNF on adolescent internalizing symptoms.

ELIGIBILITY:
Inclusion Criteria:

All participants inclusion criteria:

* Biological female
* Sufficient English fluency to complete tasks
* Co-residing at least 4 days per week

Inclusion criteria for adult participants:

* Primary caregiver for more than 50% of child's lifespan
* History of at least two adverse childhood experiences
* Biological parent of adolescent participant

Inclusion criteria for adolescents:

* Eligible for fMRI
* Body mass index between 16 and 40 (inclusive)
* Age 14-17 years

Exclusion Criteria:

Exclusion criteria for adolescent participants:

* Current or past psychiatric disorder
* Neurodevelopmental delay
* Medications influencing fMRI
* Medical conditions influencing fMRI

Min Age: 14 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Parent report of child's sex assigned at birth as "female" and current gender identity as "girl"
Enrollment: 210 (Estimated)
Dates: Start 2023-03-13 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Blood Oxygen Level-Dependent (BOLD) signal changes (brain activation) | One hour (measured during one scan session)
  Activation in the right anterior insular cortex and associated regions. We hypothesize that lower activity will indicate a better outcome.
Resting-state network activity | One year (change from first scan session to one-year follow-up)
  Brain activity during fMRI resting-state scan

SECONDARY OUTCOMES:
Depressive symptoms (change over time) | One year (change from first scan session to one-year follow-up)
  Change over time in adolescent's responses to the PROMIS (Patient Reported Outcome Measurement Information System) Pediatric Short Form Version 2 (Quinn et al., 2014). This is an 8-item scale with scores ranging from 8-40, with higher scores indicating more depressive symptoms.
Parenting behaviors (change over time) | One year (change from first scan session to one-year follow-up)
  Change over time in adolescent's responses to the Children's Report of Parent Behavior Inventory (Schludermann & Schludermann, 1988). The CRPBI has 3 subscales, each with a score range of 10-30. Interpretation/valence of the scores varies by subscale.
Emotion regulation (change over time) | One year (change from first scan session to one-year follow-up)
  Change over time in adolescent's responses to the Difficulties in Emotion Regulation Scale (Gratz & Roemer, 2008). The DERS consists of 36 items rated on a 1-5 Likert scale (scale range: 36-180). Higher scores indicate greater difficulties with emotion regulation.
Parent-adolescent interaction quality (change over time) | Two weeks
  Adolescents will complete ecological momentary assessment (EMA) measures multiple times per day over a period of two weeks and report on emotions experienced during interactions with their mother. The ratio of positive to negative interactions across the EMA period will be calculated.
Affect variability (change over time) | Two weeks
  Adolescents will complete ecological momentary assessment (EMA) measures multiple times per day over a period of two weeks and rate their current emotions at the time of the prompt. Affect variability will be quantified as the standard deviation in mean negative emotion ratings.

CONTACTS AND LOCATIONS:
Overall Officials: Kara L Kerr, PhD, Principal Investigator — Oklahoma State University
Locations (1):
- Hardesty Center for Clinical Research and Neuroscience, Tulsa, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: Undecided